CLINICAL TRIAL: NCT04083092
Title: Surveillance of Community-Associated MRSA and Treatment Outcomes of Skin and Soft Tissue Infections in the Ambulatory Setting
Brief Title: Surveillance of Community-Associated MRSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Lilly, Pediatric Infectious Disease Specialist, Children's Healthcare of Atlanta
Other Study IDs: 14-166
Record Dates: First submitted 2019-08-29; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: MRSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to obtain information from patients diagnosed with a skin and soft tissue infection (also known as an abscess or 'boil' or 'rising') and determine whether or not MRSA is present in the child's different surface skin areas or nose. We also plan to compare how these infections look in the lab, by identifying in detail parts of the germ that caused the infection or is found on the skin/nose areas

DETAILED DESCRIPTION:
Patients come into the Emergency Department for skin and soft tissue infections, which could be caused by a germ not treatable with common medications. This germ is a bacterium called methicillin-resistant Staphylococcus aureus (MRSA). MRSA is a bacterium that has become resistant to certain antibiotics. Scientists and doctors are not sure what causes individuals to develop these infections, but it is believed to be related to the bacteria that might be on a patient's skin or in their nose. Patients will be interviewed by someone from the research team to gather more details about possible risk factors related to MRSA infections. Th interview is expected to last between 10-20 minutes. Nasal (nose), axillary (armpit), throat, and around rectum swabs will be obtained by the research team as follows: Culture swabs (similar to a large Q-tip) will be inserted gently into the front half of each nostril (nare), under each arm, in the throat area, and around the perirectal area (surface skin around rectal opening) either before or after being seen by the emergency room physician. Another culture swab of the patient's skin and soft tissue infection might be taken as part of their usual care for the child's condition or a swab culture will be taken from the infection site by research personnel. A 'culture' swab is a sterile Q-tip like swab which is used to collect potential bacteria from the skin and nose, and then can be used in the laboratory to grow the bacteria collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of skin and soft tissue infections (abscesses and cellulitis)
* Patient aged >6 months and <21 years

Exclusion Criteria:

* Currently on antibiotics
* Unimmunized patients
* Pertinent co-morbid conditions (immune deficiency, underlying cardiac, skin, GI disorder)

Ages: 6 Months to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children's is the largest pediatric clinical care provider in the country. Currently, across the three hospitals (Hughes Spalding, Egleston, and Scottish Rite), there are 561 licensed beds. In 2013, CHOA managed more than 860,849 patient visits, with over 218,231 Emergency Department visits.
  Enrolled patients will be tested for colonization by CA-MRSA and CA-MSSA by standard swabbing of specified sites (nares, axilla, oropharyngeal, and perirectal areas). A culture swab will also be taken of an enrolled patient's wound infection (skin and soft tissue infection).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-07-08 (Estimated); Study Completion 2020-07-08 (Estimated)

PRIMARY OUTCOMES:
Number of children with MRSA and MSSA carriage | 1 year
  We are measuring this by swabbing 5 locations on the body of each study participant. We are swabbing the anterior nares (nostrils), under both axilla (armpits), oropharyngeal area (mouth), skin around the perirectal area, and the actual abscess wound.
Number of children with MRSA and MSSA skin and soft tissue infections | 1 year
  We are measuring this by collecting wound cultures from all children who present with skin and soft issue infections.

SECONDARY OUTCOMES:
Number of strains of MRSA and MSSA with unique genomic sequences | 1 year
  We are conducting genomic sequences. We want to understand the relationship between the different strains of MRSA and MSSA.
Percent relatedness between MRSA and MSSA protein profiles | 1 year
  Few studies have looked at the relationship between molecular characterization and treatment outcomes of children who present for skin and soft tissue infections. We will be using Matrix-assisted laser desorption ionization-time of flight (MALDI-TOF).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States